CLINICAL TRIAL: NCT02673606
Title: The Influence of Estrogen on the Fear Extinction Network in Humans-R61
Brief Title: Impact of Estrogen on Fear Extinction R61
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2007P000496
Record Dates: First submitted 2016-01-26; First posted 2016-02-04 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Fear; Fear; Examination, Phobic
MeSH Terms: interventions — Estradiol; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind placebo control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Estradiol 2mg Dose (Experimental): 2mg dose of estradiol (oral administration)
  Interventions: Drug: Estradiol 2Mg Tablet
- Estradiol 4mg Dose (Experimental): 4mg dose of estradiol (oral administration)
  Interventions: Drug: Estradiol 4Mg Tablet
- Placebo (Placebo Comparator): placebo (oral administration)
  Interventions: Drug: Placebo Pills

INTERVENTIONS:
Drug: Estradiol 2Mg Tablet — one 2 mg dose of estradiol (obtained from Estrace® Tablets, 2.0 mg estradiol tablets, USP, Warner Chilcott),
  Other Names: Estrace® Tablets
  Arms: Estradiol 2mg Dose
Drug: Estradiol 4Mg Tablet — two 2 mg pills estradiol(obtained from Estrace® Tablets, 2.0 mg estradiol tablets, USP, Warner Chilcott),
  Other Names: Estrace® Tablets
  Arms: Estradiol 4mg Dose
Drug: Placebo Pills — inactive placebo pills
  Other Names: Estrace® Tablets
  Arms: Placebo

SUMMARY:
The goal of this project is to examine how estrogen may influence the resting-state connectivity and the extinction-induced activation of the fear extinction network.

DETAILED DESCRIPTION:
The aim of the study was to examine the influence of exogenous estrogen administration on the activation of the fear extinction network in women. Functional MRI data and psychophysiological indices were collected to test the influence of estrogen on women's ability to regulate conditioned fear responses. Women underwent a 3 day experimental paradigm using classical fear conditioning. The first day was conducted outside the scanner, while days 2 and 3 were done inside the fMRI scanner and tested fear extinction learning and recall in days 2 and 3, respectively. The estrogen (or placebo) pill was given just hours before extinction learning test on day 2. No followups were conducted after women completed the 3 day study.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed (Edinburgh Inventory - Oldfield 1971).
* SCID diagnosis consistent with none, current or past history of Axis I psychiatric disorders.
* To be matched for age, gender, and years of education, as well as self-identified race/ethnicity.
* For naturally cycling female subjects, stage of menstrual cycle will be ascertained by history, and by serological measures.
* For women on oral contraceptives, we will identify those using 20mcg ethinyl, 2nd or 3rd generation, monophasic

Exclusion Criteria:

* Psychiatric, neurologic or medical condition that would interfere with study procedures or confound results, ascertained by history.
* History of seizure or significant head trauma (i.e., extended loss of consciousness, neurological sequelae, or known structural brain lesion).
* History of Axis I psychiatric diagnosis; e.g., history of substance use disorder, psychotic disorder, bipolar disorder, tic disorder, or eating disorder.
* Use of psychotropic medication within 4 weeks prior to study (within 6 weeks for fluoxetine, or other long-lived compounds; within one year for neuroleptics).
* Pregnancy (to be ruled out by urine ß-HCG).
* Metallic implants or devices contraindicating magnetic resonance imaging.
* Use of oral contraceptives or non-oral contraceptives containing estrogen and progesterone within 3 months
* History of breast cancer.
* Allergy to peanut oil.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Impact of exogenous administration of estradiol on the neural correlates of fear extinction | 3 Days
  BOLD responses during fear extinction after taking estradiol or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milad, PhD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States